CLINICAL TRIAL: NCT02457351
Title: An Open-label, Non-randomized, Phase I Study to Evaluate the Effect of Itraconazole on the Pharmacokinetics of a Single Oral Dose of Roniciclib in Patients With Advanced Solid Tumors
Brief Title: Roniciclib (BAY 1000394) Drug-Drug Interaction (DDI) Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 17616
Record Dates: First submitted 2015-05-28; First posted 2015-05-29 (Estimated); Last update posted 2016-05-23 (Estimated); Status verified 2016-05

CONDITIONS: Medical Oncology
Keywords: Phase 1; Advanced solid tumor; pan-CDK inhibitor; Drug-drug Interaction
MeSH Terms: interventions — roniciclib; Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Roniciclib + Itraconazole (Experimental): Pharmacokinetics and safety in patients with advanced solid tumor
  Interventions: Drug: Roniciclib (BAY 1000394); Drug: Itraconazole (Sporanox)

INTERVENTIONS:
Drug: Roniciclib (BAY 1000394) — Part 1 of Cycle 1 Cycle 1 Day 1: Single dose 2.5 mg Cycle 1 Day 6: Single dose 2.5 mg Part 2 of Cycle 1 Cycle 1 Day 1: Single dose 2.5 or 5 mg (based on Part 1 data) Cycle 1 Day 6: Single dose 2.5 or 5 mg (based on part 1 data)
  Part 1 & Part 2
  Cycle 2 and subsequent 21-day cycles:
  Day 1-3 of each cycle: 5 mg bid Day 4-7 of each cycle: no dose
Drug: Itraconazole (Sporanox) — Part 1 & Part 2 of Cycle 1 Cycle 1 Day 4: 200 mg bid Cycle 1 Day 5-11: 200 mg qd

SUMMARY:
To evaluate the effect of itraconazole, a strong CYP3A4 inhibitor, on the pharmacokinetics of roniciclib in cancer patients.

To assess safety and tolerability of roniciclib dosing when administered with and without itraconazole in cancer patients

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients ≥ 18 years of age with histological or cytological confirmed advanced solid tumors refractory to, or not able to tolerate to any standard therapy, have no standard therapy available, or subjects must have actively refused any treatment which would be regarded standard, and / or if in the judgment of the investigator, experimental treatment is clinically and ethically acceptable.
* Adequate liver, renal and bone-marrow functions as assessed by laboratory values.
* ECOG Performance Status of 0 - 2 and life expectancy of at least 12 weeks.
* Subject with a history of hypertension should be on a stable anti-hypertensive treatment for more than 7 days prior to the first dose of study drug.

Exclusion Criteria:

Medical and surgical history:

* Previous deep vein thrombosis (within the last 6 months), arterial thrombotic events (including strokes), or pulmonary embolism.
* History of cardiac disease: congestive heart failure, angina (within past 6 months prior to study entry), myocardial infarction, or cardiac arrhythmias requiring anti-arrhythmic therapy (beta blockers or digoxin are permitted).
* Uncontrolled hypertension (systolic blood pressure >150 mmHg or diastolic blood pressure >90 mmHg despite optimal medical management)
* Moderate or severe hepatic impairment, i.e. Child-Pugh class B or C. History of human immunodeficiency virus (HIV) infection or chronic hepatitis B or C
* Active clinically serious infections of Common Terminology Criteria for Adverse Events (CTCAE, v. 4.03) > Grade 2.
* Symptomatic metastatic brain or meningeal tumors unless the subject is >3 months from definitive therapy, has no evidence of tumor growth on an imaging study within 4 weeks prior to study entry, and is clinically stable with respect to the tumor at the time of study entry.
* Seizure disorder requiring therapy (such as steroids or anti-epileptics).
* History of organ allograft.
* Use of strong inhibitors and/or inducers of CYP3A4 in the 14 days before study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2015-07; Primary Completion 2016-02 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Maximum observed drug concentration (Cmax) of roniciclib on Cycle 1 Day 1 (without itraconazole) | Cycle 1 Day 1: pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 24, 48 and 72 hours after dosing
Area under the concentration vs. time curve from zero to infinity (AUC) of roniciclib on Cycle 1 Day 1 (without itraconazole) | Cycle 1 Day 1: pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 24, 48 and 72 hours after dosing
Maximum observed drug concentration (Cmax) of roniciclib on Cycle 1 Day 6 (with itraconazole) | Cycle 1 Day 6: pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 24, 48, 72, 96 and 120 hours after dosing
Area under the concentration vs. time curve from zero to infinity (AUC) of roniciclib on Cycle 1 Day 6 (with itraconazole) | Cycle 1 Day 6: pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 24, 48, 72, 96 and 120 hours after dosing

SECONDARY OUTCOMES:
Collection of Adverse events as a measure of safety and tolerability of roniciclib dosing when administered with and without itraconazole | up to 15 months
Laboratory analyses to assess safety and tolerability of roniciclib dosing when administered with and without itraconazole | up to 15 months
  Complete blood count, Complete chemistry panel, Coagulation panel, Virology, Urinalysis, Pregnancy test
Monitoring of vital signs to assess safety and tolerability of roniciclib dosing when administered with and without itraconazole | up to 15 months
East Coast Oncology Group (ECOG) performance status to assess safety and tolerability of roniciclib dosing when administered with and without itraconazole | up to 15 months
Electrocardiogram (12 lead ECG) readings to assess safety and tolerability of roniciclib dosing when administered with and without itraconazole | up to 15 months
Physical examination to assess safety and tolerability of roniciclib dosing when administered with and without itraconazole | up to 15 months
Maximum observed drug concentration (Cmax) of roniciclib after a light meal on Cycle 1 Day -2 (without itraconazole) | Cycle 1 Day -2: pre-dose, 0.5, 1, 2, 3, 4, 6, 8, and 24 hours after dosing
Area under the concentration vs. time curve from zero to 24 hr (AUC) of roniciclib after a light meal on Cycle 1 Day -2 (without itraconazole) | Cycle 1 Day -2: pre-dose, 0.5, 1, 2, 3, 4, 6, 8, and 24 hours after dosing

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (4):
- Canada (4):
  - Edmonton, Alberta
  - Hamilton, Ontario
  - London, Ontario
  - Montreal, Quebec